CLINICAL TRIAL: NCT06327958
Title: THE EFFECTS OF DIRECT AND INDIRECT LARYNGOSCOPY ON CORMACK-LEHANE AND POGO SCORES IN THE LARYNGOSCOPY TRAINING OF MEDICAL STUDENTS: A SIMULATION STUDY
Brief Title: THE EFFECTS OF DIRECT AND INDIRECT LARYNGOSCOPY ON CORMACK-LEHANE AND POGO SCORES
Status: Completed | Type: Observational
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Gamze Küçükosman, Associate Professor, Zonguldak Bulent Ecevit University
Other Study IDs: protocol Number: 2021/21
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2022-06

CONDITIONS: Being a 5th Year Student at the Faculty of Medicine; No Previous Laryngoscopy Experience
Keywords: Cormack-Lehane; percentage of glottic opening (POGO) score; medical students.; manikin study

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: McGRATH-MAC Videolaryngoscope,: Cormack-Lehane (C&L) and percentage of glottic opening (POGO) scores in the airway management training of medical students.
  Interventions: Other: Cormack-Lehane (C&L); Other: POGO score
- Group 2: C-MAC Videolaryngoscopy: Cormack-Lehane (C&L) and percentage of glottic opening (POGO) scores in the airway management training of medical students.
  Interventions: Other: Cormack-Lehane (C&L); Other: POGO score
- Group 3: Macintosh Laryngoscope.: Cormack-Lehane (C&L) and percentage of glottic opening (POGO) scores in the airway management training of medical students.
  Interventions: Other: Cormack-Lehane (C&L); Other: POGO score

INTERVENTIONS:
Other: Cormack-Lehane (C&L) — There is no distinguishing feature of the C&L and POGO scores required to provide the best laryngoscopic view from other interventions in this or any other clinical trial.
Other: POGO score — There is no distinguishing feature of the C&L and POGO scores required to provide the best laryngoscopic view from other interventions in this or any other clinical trial.

SUMMARY:
Direct laryngoscopy (DL) is a conventional and highly difficult method that is used in endotracheal intubation (ETI) training. Today, the usage of video-laryngoscopes (VLs) to teach airway management to inexperienced healthcare personnel is a prevalent practice. In ETI training, it is recommended to train students on simulators before allowing them direct access to patients.

ELIGIBILITY:
Inclusion Criteria:

* Students who were informed,
* whose informed consent was received were invited to participate in the study

Exclusion Criteria:

* Students who were experienced in laryngoscopy,
* those who had received relevant training,
* those who had watched videos on the subject,
* those who refused to participate were excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The population was determined as students who participated in anesthesiology internships in the 2021-2022 academic year.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
The percentage of glottic opening (POGO) scores in the airway management training of medical students. | September 2021-June 2022

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bülent Ecevit University, Zonguldak, Kozlu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No